CLINICAL TRIAL: NCT03282006
Title: The Efficacy and Safety of Pivmecillinam in Treating Bacteriemic Urosepsis Caused by E.Coli
Brief Title: Treating Pyelonephritis an Urosepsis With Pivmecillinam
Acronym: MePUr
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sykehuset i Vestfold HF (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Tore Stenstad, MD, PhD, Sykehuset i Vestfold HF
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-000984-18
Record Dates: First submitted 2017-04-25; First posted 2017-09-13 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Pyelonephritis; Urinary Tract Infections
Keywords: Pivmecillinam
MeSH Terms: conditions — Pyelonephritis; Urinary Tract Infections | interventions — Amdinocillin Pivoxil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pivmecillinam (Experimental): Patients treated with pivmecillinam
  Interventions: Drug: pivmecillinam

INTERVENTIONS:
Drug: pivmecillinam — Oral treatment of bacteremic pyelonephritis following standard initial parenteral treatment
  Other Names: Selexid, Penomax

SUMMARY:
Febrile urinary tract infections and urosepsis are common and potentially serious infections that require effective antimicrobial treatment. The duration of parenteral treatment depends on oral alternatives. These alternatives are few and due to antimicrobial resistance, quinolones are "standard of care". The increased use of quinolones is concerning because of its negative ecological aspects and it is confirmed an increasing incidence of resistant E.coli to quinolones in Norwegian isolates.

Pivmecillinam is an antibiotic with high susceptibility to E.coli but the evidence for treating febrile urinary tract infections is insufficient. This trial will investigate the efficacy and safety of pivmecillinam in treating pyelonephritis and urosepsis caused by E.coli.

The hypothesis is that urosepsis can safely be treated with pivmecillinam when it is given after 2-3 days with empirical i.v. antibiotics.

DETAILED DESCRIPTION:
This trial will be conducted at Vestfold Hospital, Norway, and is a prospective observational study with intention to treat. Participants will be consecutively included among hospitalized patients suffering from urosepsis - see eligibility criteria. After 3 days with parenteral antibiotics, when clinical improvement and absence of fever/leukocytosis is confirmed, the participants will start on pivmecillinam 400mg four times daily and be discharged. Pivmecillinam is to be taken for one week. The participants will be contacted by phone on day 4, 10 and 33 (days after admission). On day 17 (test of cure, TOC) they will meet for physical examination. They will report symptom score (standardized schema) on day 0, and 17. Urine samples will be collected on day 10 and 17. Blood samples on day 17. All data will be stored anonymously. The trial will be monitored by extern resources.

ELIGIBILITY:
Inclusion Criteria:

* E.coli in blood culture
* AND identical isolate in urine sample (>= 1.000 CFU) OR relevant clinical signs of UTI

Exclusion Criteria:

* Bacterial infection origin from another organ (e.g. pneumonia)
* Severe sepsis with multiorgan failure
* Perinephritic abscess
* Pyonephrosis requiring drainage
* Allergy to pivmecillinam
* E.coli isolate resistant to pivmecillinam
* Pregnancy/breastfeeding
* Severe neutropenia
* Prostatitis
* Severe kidney failure (eGFR<15 ml/min)
* Using valproate

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2020-04-21 (Actual); Study Completion 2020-04-21 (Actual)

PRIMARY OUTCOMES:
Clinical efficacy | Day 17
  Defined as abscence of fever, no need for other antibiotics than prescribed and improvement of symptoms (self-reported improvement and EQ 5D VAS-scale).

SECONDARY OUTCOMES:
C-reactive protein-level (CRP) | Day 17
  Compare CRP-level on day 0 with day 17.
Readmission due to urinary tract infection (UTI) | Day 33
  Check if participants are readmitted due to UTI.
Readmission - any cause | Day 33
  Check if participants have been readmitted to hospital
Adverse effects | Day 33
  Registrate frequency of rash/skin problems, abdominal pain, clostridium difficile associated diarrhea
Microbial efficacy | Day 17
  Defined as <1.000 CFU E.coli in urine

CONTACTS AND LOCATIONS:
Overall Officials: Tore Stenstad, MD, PhD, Principal Investigator — The Hospital of Vestfold
Locations (1):
- Vestfold Hospital Trust, Tønsberg, Vestfold, Norway

REFERENCES:
- [Derived] Hansen BA, Grude N, Lindbaek M, Stenstad T. The efficacy of pivmecillinam in oral step-down treatment in hospitalised patients with E. coli bacteremic urinary tract infection; a single-arm, uncontrolled treatment study. BMC Infect Dis. 2022 May 19;22(1):478. doi: 10.1186/s12879-022-07463-7. PMID 35590284